CLINICAL TRIAL: NCT01393132
Title: Comparative Study of Thymosin Beta 4 Eye Drops or Vehicle in the Treatment of Patients With Ocular Surface Defects Due to Severe Dry Eye
Brief Title: Comparative Study of Thymosin Beta 4 Eye Drops vs. Vehicle in the Treatment of Severe Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michigan Cornea Consultants, PC (Other)
Collaborators: Kresge Eye Institute (Other)
Responsible Party: Principal Investigator, Steven P. Dunn, M.D., Principal Investigator, Michigan Cornea Consultants, PC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1003008179
Record Dates: First submitted 2011-07-07; First posted 2011-07-13 (Estimated); Results first posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Dry Eye; Sjogren's Syndrome; Graft vs. Host Disease
Keywords: Dry Eye; Sjogren's Syndrome; Graft vs. Host Disease; Rheumatoid arthritis; Systemic lupus erythematosus; Scleroderma
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome; Graft vs Host Disease; Arthritis, Rheumatoid; Lupus Erythematosus, Systemic; Scleroderma, Diffuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thymosin Beta 4 eye drops (Experimental): It is a preservative-free, sterile eye drop solution containing Tβ4 for direct instillation into each eye, six times daily for 28 days
  Interventions: Drug: Thymosin Beta 4 eye drops
- Vehicle Control (Placebo Comparator): It is composed of the same excipients as RGN-259 but does not contain Tβ4 for direct instillation into each eye, six times daily for 28 days.
  Interventions: Drug: Vehicle Control

INTERVENTIONS:
Drug: Thymosin Beta 4 eye drops — Patients will be randomized and will receive the same eye drops the Thymosin Beta 4.
  Other Names: Tβ4
  Arms: Thymosin Beta 4 eye drops
Drug: Vehicle Control — Patients will be randomized and will receive the same eye drops without the Thymosin Beta 4.
  Other Names: Vehicle
  Arms: Vehicle Control

SUMMARY:
Severe dry eye is a debilitating ocular disease resulting in loss of vision, reduced day-to-day function and significant discomfort. Tear substitutes are an important part of the treatment of all patients, however, even with aggressive us, the corneal(ocular)surface often remains very irregular due to poor surface healing.

The agent being evaluated in this study, Thymosin Beta 4, promotes healing of the corneal surface and has been studied in patients with recalcitrant corneal ulcers and erosions with significant success (Arch Ophthalmol. 2010;128(5):636-638., Ann of the NY Acad of Sci, May, 2010).

The study hypothesis is that Thymosin Beta 4, in its role as a modulator of corneal surface healing, may be able to promote healing of the corneal surface allowing for more conventional modalities to take over and maintain a smooth and regular ocular surface. The investigators hope to be able to demonstrate an improvement in visual acuity, surface healing and a reduction in dry-eye related symptoms.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* Schirmers of < 5 mm at 5 minutes
* TFBUT: less than 10 seconds
* Corneal staining of >3 of 15: conjunctival staining of >3 of 18
* Ocular Surface Disease Index of > 50
* Presumed best corrected vision of 20/60 or better

Exclusion Criteria:

* Acute or inflammatory corneal disease
* Pregnancy or lactation
* Monocular status
* Punctal occlusion within 30 days
* Ocular surgery within 3 months
* Corneal thinning of >50%
* Active corneal infection
* History of ocular malignancy
* Retinal neovascularization
* Current use of topical cyclosporin A

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Dunn, M.D., Principal Investigator — Michigan Cornea Consultants, P.C.
Locations (1):
- Michigan Cornea Consultants, P.C., Southfield, Michigan, United States

REFERENCES:
- [Derived] Sosne G, Dunn SP, Kim C. Thymosin beta4 significantly improves signs and symptoms of severe dry eye in a phase 2 randomized trial. Cornea. 2015 May;34(5):491-6. doi: 10.1097/ICO.0000000000000379. PMID 25826322

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Details The study took place at Kresge Eye Institute by Dr. Gabriel Sosne, and at Michigan Cornea Consultants, P.C. by Dr. Steven P. Dunn,
  The first subject was screened on Mar.2011 and the last subject last visit to the clinic was on Dec.2012
Pre-assignment Details: Pre-assignment Details:
  Subjects were evaluated upon entering the study after a two week washout period.
Groups:
- Thymosin: Arm/Group * Reporting Groups Definition: Arms or comparison groups in a trial
  Description Placebo : A preservative-free, sterile eye drop solution not including Tβ4 for direct instillation into each eye, six times daily for 28 days.
  Thymosin beta 4 : A preservative-free, sterile eye drop solution containing 0.1% (w/w) Tβ4 for direct instillation into each eye, six times daily for 28 days.
  Period Title * Participant Flow: Overall Study
  Placebo Thymosin Beta 4 Started 3 6 Completed 3 6
- Placebo: Arm/Group * Reporting Groups Definition: Arms or comparison groups in a trial
  Description Placebo : A preservative-free, sterile eye drop solution not including Tβ4 for direct instillation into each eye, six times daily for 28 days.
Period: Overall Study
Arm/Group | Thymosin | Placebo
Started | 6 | 3
Completed | 6 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Thymosin; Placebo: Comparison
  Thymosin Beta 4 eye drops vs. vehicle: Patients will be randomized and will receive either Thymosin Beta 4 eye drops or the same eye drops without the Thymosin Beta 4.
- Total: Total of all reporting groups
Arm/Group | Thymosin | Placebo | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 7
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.2 (11.6) | 63.7 (6.65) | 57.33 (11.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Safety
Description: Sum of adverse events observed at Day 1, Day 14, Day 28 and Day 56. Measurable by Intra-ocular pressure (IOP) by applanation tonometry, Complete ophthalmologic evaluation including fundoscopy, An adverse event (baseline and all subsequent study visits).
Time Frame: Day 1, Day 14, Day 28 and Day 56
Measure: Number; unit: event
Groups:
- Thymosin: Thymosin beta 4 : A preservative-free, sterile eye drop solution containing 0.1% (w/w) Tβ4 for direct instillation into each eye, six times daily for 28 days.
- Placebo: Placebo : A preservative-free, sterile eye drop solution not including Tβ4 for direct instillation into each eye, six times daily for 28 days
Arm/Group | Thymosin | Placebo
Number analyzed (Participants) | 6 | 3
event | 0 | 0

2. Secondary Outcome: Corneal Fluorescein Staining
Description: Ocular surface irregularity as measured by Slit Lamp Examination (SLE) with fluorescein dye staining of the cornea at days 56 (+28 day follow up).
  The scale used to determine the difference in corneal fluorescein staining is the Oxford scale. (The Oxford Scale measures corneal fluorescein staining) Corneal staining type was assessed by the investigator for each of 5 regions of the cornea, i.e., four quadrants plus central. The five regions were summed, for a maximum score of 25. A higher score represents greater disability.
Time Frame: Days 56 (+28 day follow up)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thymosin | Placebo
Number analyzed (Participants) | 6 | 3
units on a scale | 4.5 (3.406) | 11.0 (4.927)
Statistical Analysis 1: Comparison: Thymosin vs Placebo; Comparison of fluorescein staining score between the placebo and Thymosin beta 4 groups; Test type: Superiority or Other; p = 0.0108, t-test, 2 sided

3. Secondary Outcome: Ocular Discomfort Index
Description: Dry eye causes ocular discomfort, which is measured using a Ocular Surface Disease Index at 56 day (+28 day followup).
  (Symptomatic improvement using the validated Ocular Surface Disease Index (OSDI).
  The OSDI is a questionnaire that consists of 12 questions about ocular irritation and the effect of dry eye on vision.
  For every question, participants check a score between 0 and 4, where 0 equals "none of the time" and 4 equals "all of the time.
  OSDI scores are calculated according to: OSDI = [(sum of scores for all questions answered)*100] / [(total number of questions answered)*4].
  The OSDI is scored on a scale of 0 to 100, with higher scores representing greater disability.
Time Frame: Days 56 (+28 day follow up)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thymosin | Placebo
Number analyzed (Participants) | 6 | 3
units on a scale | 45.625 (17.780) | 67.233 (15.658)
Statistical Analysis 1: Comparison: Thymosin vs Placebo; Comparison of Ocular Discomfort Index score between the placebo and Thymosin beta 4 groups; Test type: Superiority or Other; p = 0.0141, t-test, 2 sided

4. Secondary Outcome: Tear Film Break up Time
Description: Tear film break up time (TFBUT) was measured to evaluating the quality of tear at 56 day (+28 day follow up).
  The tear film break-up time is defined as the interval between the last complete blink and the first appearance of a dry spot, or disruption in the tear film.
  Range : >10 seconds is thought to be normal, <5 seconds low (with high likelihood of dry eye symptoms).
Time Frame: Days 56 (+28 day follow up)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Thymosin | Placebo
Number analyzed (Participants) | 6 | 3
seconds | 5.550 (2.302) | 2.848 (1.137)
Statistical Analysis 1: Comparison: Thymosin vs Placebo; Comparison of Tear Film Break up Time between the placebo and Thymosin beta 4 groups; Test type: Superiority or Other; p = 0.0162, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 56 days
Groups:
- Thymosin Beta 4: Thymosin beta 4 : A preservative-free, sterile eye drop solution containing 0.1% (w/w) Tβ4 for direct instillation into each eye, six times daily for 28 days.
- Placebo: : A preservative-free, sterile eye drop solution not including Tβ4 for direct instillation into each eye, six times daily for 28 days
Arm/Group | Thymosin Beta 4 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 0/6 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No